CLINICAL TRIAL: NCT05880368
Title: Partnership in Resilience for Medication Safety
Brief Title: Partnership in Resilience for Medication Safety (PROMIS)
Acronym: PROMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-0439
Record Dates: First submitted 2023-05-11; First posted 2023-05-30 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Patient Engagement; Patient Empowerment; Patient Activation
Keywords: Medication safety; Primary care
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: Stepped wedge with a parallel control arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient partnership tool (Experimental): Study participants as patients visiting primary care providers in the clinics using the study patient engagement tools aimed to reduce preventable adverse drug events.
  Interventions: Other: Patient partnership tools
- Control (No Intervention): Study participants as patients visiting primary care providers in the clinics without the study patient engagement tools.

INTERVENTIONS:
Other: Patient partnership tools — The intervention consists of two patient partnership tools: (1) a one-page 'visit prep guide' given to relevant patients by clinic staff before seeing the primary care provider, with the intention to improve communication and shared decision-making; and (2) a series of short educational videos that clinic staff can encourage patients to watch. The interventions will be included in the workflow of the clinics during the intervention periods (i.e., clinics either do not use the intervention or use them for all relevant patients depending on study period).
  Arms: Patient partnership tool

SUMMARY:
The trial is to assess the impact of two patient partnership tools: (1) a one-page 'visit prep guide' given to relevant patients by clinic staff before seeing the provider, with the intention to improve communication and shared decision-making; and (2) a series of short educational videos that clinic staff can encourage patients to watch.

DETAILED DESCRIPTION:
Preventable patient harms from medications are significant threats to patient safety in ambulatory and community settings and contributed 700,000 emergency department visits each year. More than a third of community-dwelling 65 years or older adults take 5 or more prescription medications. In ambulatory and community settings, more so than in inpatient settings, medication safety is shaped by interactions among patient/caregivers and different professionals across locations. We developed a set of patient partnership tools to encourage and empower patients to make use of their office visits through setting expectations of information sharing, learning basics of medication self-management, and working with community pharmacy resources. The trial will be conducted at private and safety-net primary care clinics to assess the impact of the partnership tools: 1) a one-page 'visit prep guide' given to relevant patients by clinic staff before seeing the provider, with the intention to improve communication and shared decision-making; and (2) a series of short educational videos that clinic staff can encourage patients to watch. A step-wedge design will be used, with medication use self-efficacy as the primary outcome, as measured by a validated tool. Secondary outcomes are issues identified by medication review.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling (e.g., not in skilled nursing facilities)
* Age 50 years or older
* Taking 5 or more medications
* English or Spanish speaking

Exclusion Criteria:

* Non-English and non-Spanish speaking
* Impaired decision making capacity
* Non-consenting

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Medication use and self-efficacy | Within 4 hours after primary care visit (one time assessment)
  Medication use and self-efficacy, which is a validated 8-item, 4-point Likert scale survey with a score range of 8-32 and higher indicating higher self-efficacy. The items are: (1) It is easy for me to take my medicine on time, (2) It is easy to remember to take all my medicines, (3) It is easy for me to set a schedule to take my medicines each day, (4) It is easy for me to take my medicines each day, (5) It is easy for me to ask my pharmacist questions about my medicine, (6) It is easy for me to understand my pharmacist's instructions for my medicine, (7) It is easy for me to understand instructions on medicine bottles, (8) It is easy for me to get all the information I need about my medicine.

SECONDARY OUTCOMES:
Medication regimen problems | Within 4 hours after primary care visit (one time assessment)
  The number of medication regimen problems identified by the provider during the visit, using a medication review form, with higher number of problems indicating higher risks for medication regimen problems. Different types of regimen problems, such as unintentional duplication, will be countered and added.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Xiao, PhD, Principal Investigator — University of Texas at Arlington
Locations (2):
- United States (2):
  - Texas Health Care, Fort Worth, Texas
  - John Peter Smith Health, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect patient privacy.

REFERENCES:
- [Background] Cameron KA, Ross EL, Clayman ML, Bergeron AR, Federman AD, Bailey SC, Davis TC, Wolf MS. Measuring patients' self-efficacy in understanding and using prescription medication. Patient Educ Couns. 2010 Sep;80(3):372-6. doi: 10.1016/j.pec.2010.06.029. Epub 2010 Jul 21. PMID 20650594
- [Background] Brega AG, Barnard J, Mabachi NM, et al. AHRQ Health Literacy Universal Precautions Toolkit, Second Edition. Rockville, MD: AHRQ Publication No. 15-0023-EF;2015
- [Derived] Xiao Y, Fulda KG, Young RA, Hendrix ZN, Daniel KM, Chen KY, Zhou Y, Roye JL, Kosmari L, Wilson J, Espinoza AM, Sutcliffe KM, Pitts SI, Arbaje AI, Chui MA, Blair S, Sloan D, Jackson M, Gurses AP. Patient Partnership Tools to Support Medication Safety in Community-Dwelling Older Adults: Protocol for a Nonrandomized Stepped Wedge Clinical Trial. JMIR Res Protoc. 2024 Apr 29;13:e57878. doi: 10.2196/57878. PMID 38684080

DOCUMENTS (2):
  • Informed Consent Form: Patient engagement survey consent form (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT05880368/ICF_000.pdf
  • Informed Consent Form: Provider consent form (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT05880368/ICF_001.pdf